CLINICAL TRIAL: NCT07397403
Title: The Efficacy of Doxycycline Post Exposure Prophylaxis for Preventing Sexually Transmitted Diseases (Gonorrhea, Chlamydia, Syphilis) Among Men Who Have Sex With Men in Bangkok, Thailand.
Brief Title: The Efficacy of Doxycycline Post Exposure Prophylaxis for Preventing STIs Among MSM in Bangkok, Thailand.
Acronym: ThaiDoxyPEP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bangrak STIs Center (Other Government)
Collaborators: Mahidol University (Other)
Responsible Party: Principal Investigator, Rossaphorn Kittiyaowamarn, Chief of Bangrak STIs Center, Bangrak STIs Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1/2568
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-10

CONDITIONS: Syphilis Infection; Gonorrhea; Chlamydia
Keywords: DoxyPEP; MSM; Syphilis; gonorrhea; Chlamydia; Prevention
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections; Syphilis | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized controlled trial (RCT). Participants will be randomly assigned to either the intervention group or the control group in a 2:1 ratio using simple randomization.
  The intervention group will receive doxycycline for the prevention of sexually transmitted infections (gonorrhea, chlamydia, and syphilis) for a period of 3 months. The control group will receive standard-of-care services and a brief educational session on sexually transmitted infection prevention at the start of the study.
  All participants will be tested for bacterial sexually transmitted infections (syphilis, gonorrhea, and chlamydia) at baseline and again at the end of the study after completing 12 weeks of follow-up.
  Before randomization, eligible participants will complete a questionnaire assessing knowledge, attitudes, and preventive behaviors related to sexually transmitted infections. In-depth interviews will also be conducted among men who have sex with men (MSM) at risk due
Masking Description: Labotatory staffs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DoxyPEP arm (Experimental): Participants will receive DoxyPEP for STIs prophylaxis in this arm
  Interventions: Drug: Doxycycline (200mg/day)
- Control arm (No Intervention): Participants will receive standard STIs prevention

INTERVENTIONS:
Drug: Doxycycline (200mg/day) — Doxycycline 200 mg single dose after unprotected sex within 24-72 hours
  Arms: DoxyPEP arm

SUMMARY:
The objective of this research is to evaluate the efficacy and safety of doxycycline in MSM for preventing sexually transmitted infections (gonorrhea, chlamydia, and syphilis) in Thailand

Participation in this study will last approximately 12 weeks and will include 2-3 clinic visits, along with 10-11 follow-up phone contacts over a period of 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

Biological male, aged not over 60 years

Thai nationality

Able to read, communicate, and understand the Thai language

Men who have sex with men (MSM), aged 18 years or older and not over 60 years

Having at least one of the following risk factors:

A history of condomless sex, or condom failure (breakage, leakage, or slippage), via any sexual route with at least two sexual partners within the past 3 months

A diagnosis of gonorrhea, chlamydia, or syphilis within the past 6 months

Current use of HIV pre-exposure prophylaxis (PrEP)

Willing and able to participate in study procedures (e.g., able to return to the clinic for scheduled testing for gonorrhea, chlamydia, and syphilis; able to complete doxycycline use records; and able to receive follow-up phone calls from the research team)

Willing and able to provide written informed consent to participate in the study

-

Exclusion Criteria:

* History of allergy to tetracycline-class antibiotics

Diagnosed with syphilis and not yet treated, or currently receiving treatment with benzathine penicillin G or doxycycline

Receipt of benzathine penicillin G within the past 12 weeks

Prior receipt of a gonorrhea vaccine

Current use of medications or products that may interact with doxycycline, including:

Vitamin A derivatives (e.g., isotretinoin, acitretin)

Antiepileptic drugs (e.g., phenytoin, carbamazepine, phenobarbital)

Immunosuppressive agents (e.g., methotrexate)

Medications for heart failure or cardiac arrhythmias (e.g., digoxin)

Anticoagulants (e.g., warfarin)

Use of oral or injectable medications that affect blood cells, such as anticancer drugs, chemotherapy, systemic corticosteroids, or targeted therapies

History of renal impairment (eGFR < 60 mL/min/1.73 m²) or hepatic impairment (AST or ALT > 3 times the upper limit of normal)

Uncontrolled or unstable underlying diseases, such as hematologic disorders, cancer, autoimmune diseases, or neurological disorders

Severe medical or psychiatric conditions that, in the investigator's judgment, may increase study-related risk or impair the participant's ability to provide informed consent

Alcohol dependence (inability to control alcohol consumption, withdrawal symptoms upon reduction or cessation, or continued use despite harm) or illicit drug dependence (regular, uncontrolled use) within the past 12 months prior to enrollment, which may affect doxycycline use for STI prevention

Previous participation in this study with prior randomization

Ages: 18 Days to 60 Days | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Men who have sex with men
Enrollment: 400 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of doxycycline in preventing sexually transmitted infections (gonorrhea, chlamydia, and syphilis) among men who have sex with men in Thailand. | 12 weeks
  Measure the proportion of participants who test positive by NAAT for gonorrhea or chlamydia at any anatomical site (genital, pharyngeal, or rectal), or who are diagnosed with syphilis during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Rossaphorn KITTIYAOWAMARN, MD, Principal Investigator — Bangrak STIs Center
Locations (1):
- Bangrak STIs Center, Sathorn, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be publicly shared due to ethical and legal considerations. The study involves sensitive sexual health information from key populations, and even de-identified datasets may carry a risk of re-identification. Data sharing is also subject to Thai data protection regulations and the conditions approved by the institutional ethics committee and participant informed consent.

REFERENCES:
- [Background] Frederiks WM, Kummerlin IP, Bosch KS, Vreeling-Sindelarova H, Jonker A, Van Noorden CJ. NADPH production by the pentose phosphate pathway in the zona fasciculata of rat adrenal gland. J Histochem Cytochem. 2007 Sep;55(9):975-80. doi: 10.1369/jhc.7A7222.2007. Epub 2007 May 28. PMID 17533217
- [Background] Ren Z, Zhang P, Wang H, Wang H. Qualitative research investigating the mental health care service gap in Chinese burn injury patients. BMC Health Serv Res. 2018 Nov 28;18(1):902. doi: 10.1186/s12913-018-3724-3. PMID 30486854
- [Background] Liu Q, Tong D, Yuan W, Liu G, Yuan G, Lan W, Zhang D, Zhang J, Huang Z, Zhang Y, Jiang J. Different RET gene mutation-induced multiple endocrine neoplasia type 2A in 3 Chinese families. Medicine (Baltimore). 2017 Jan;96(3):e5967. doi: 10.1097/MD.0000000000005967. PMID 28099363
- [Background] Peyriere H, Makinson A, Marchandin H, Reynes J. Doxycycline in the management of sexually transmitted infections. J Antimicrob Chemother. 2018 Mar 1;73(3):553-563. doi: 10.1093/jac/dkx420. PMID 29182717
- [Result] Stewart J, Oware K, Donnell D, Violette LR, Odoyo J, Soge OO, Scoville CW, Omollo V, Mogaka FO, Sesay FA, McClelland RS, Spinelli M, Gandhi M, Bukusi EA, Baeten JM; dPEP Kenya Study Team. Doxycycline Prophylaxis to Prevent Sexually Transmitted Infections in Women. N Engl J Med. 2023 Dec 21;389(25):2331-2340. doi: 10.1056/NEJMoa2304007. PMID 38118022
- [Result] Molina JM, Bercot B, Assoumou L, Rubenstein E, Algarte-Genin M, Pialoux G, Katlama C, Surgers L, Bebear C, Dupin N, Ouattara M, Slama L, Pavie J, Duvivier C, Loze B, Goldwirt L, Gibowski S, Ollivier M, Ghosn J, Costagliola D; ANRS 174 DOXYVAC Study Group. Doxycycline prophylaxis and meningococcal group B vaccine to prevent bacterial sexually transmitted infections in France (ANRS 174 DOXYVAC): a multicentre, open-label, randomised trial with a 2 x 2 factorial design. Lancet Infect Dis. 2024 Oct;24(10):1093-1104. doi: 10.1016/S1473-3099(24)00236-6. Epub 2024 May 23. PMID 38797183
- [Result] Luetkemeyer AF, Donnell D, Dombrowski JC, Cohen S, Grabow C, Brown CE, Malinski C, Perkins R, Nasser M, Lopez C, Vittinghoff E, Buchbinder SP, Scott H, Charlebois ED, Havlir DV, Soge OO, Celum C; DoxyPEP Study Team. Postexposure Doxycycline to Prevent Bacterial Sexually Transmitted Infections. N Engl J Med. 2023 Apr 6;388(14):1296-1306. doi: 10.1056/NEJMoa2211934. PMID 37018493
- [Result] Molina JM, Charreau I, Chidiac C, Pialoux G, Cua E, Delaugerre C, Capitant C, Rojas-Castro D, Fonsart J, Bercot B, Bebear C, Cotte L, Robineau O, Raffi F, Charbonneau P, Aslan A, Chas J, Niedbalski L, Spire B, Sagaon-Teyssier L, Carette D, Mestre SL, Dore V, Meyer L; ANRS IPERGAY Study Group. Post-exposure prophylaxis with doxycycline to prevent sexually transmitted infections in men who have sex with men: an open-label randomised substudy of the ANRS IPERGAY trial. Lancet Infect Dis. 2018 Mar;18(3):308-317. doi: 10.1016/S1473-3099(17)30725-9. Epub 2017 Dec 8. PMID 29229440
- [Result] Nanthaprut P, Manojai N, Chanlearn P, Mattawanon N, Chiawkhun P, Homkham N, Traisathit P. Comparison of HIV-Positive Incidence Among Transgender Women and Men Who Have Sex with Men at Stand-Alone and Mobile Voluntary Counseling and Testing Facilities in Chiang Mai Province, Thailand. AIDS Patient Care STDS. 2021 Apr;35(4):116-125. doi: 10.1089/apc.2020.0258. PMID 33835852
- [Result] Chen JS, Levintow SN, Tran HV, Sripaipan T, Nguyen MX, Nguyen SM, Miller WC, Go VF, Giang LM. HIV and STI prevalence and testing history among men who have sex with men in Hanoi, Vietnam. Int J STD AIDS. 2022 Feb;33(2):193-201. doi: 10.1177/09564624211060185. Epub 2021 Dec 1. PMID 34852691
- [Result] Nguyen TV, Tran HP, Khuu NV, Nguyen PD, Le TN, Hoang CD, Tran T, Le TQ, Pham QD, Phan LT. Increases in both HIV and syphilis among men who have sex with men in Vietnam: Urgent need for comprehensive responses. Int J STD AIDS. 2021 Dec;32(14):1298-1307. doi: 10.1177/09564624211036421. Epub 2021 Aug 14. PMID 34392717
- [Result] Johnston LG, Soe P, Widihastuti AS, Camellia A, Putri TA, Rakhmat FF, Nurwandani RA, Prabhu SM, Sulaiman N, Pronyk PM. Alarmingly High HIV Prevalence Among Adolescent and Young Men Who have Sex with Men (MSM) in Urban Indonesia. AIDS Behav. 2021 Nov;25(11):3687-3694. doi: 10.1007/s10461-021-03347-0. Epub 2021 Jun 18. PMID 34143341
- See also: Sexually transmitted infections (STIs) [Internet]. Who.int. [cited 2024 Sep 24]. — https://www.who.int/news-room/fact-sheets/detail/sexually-transmitted-infections-(stis)
- See also: Center for Disease Control and Prevention. Sexually transmitted infections (STIs). [cited 2024 Sep 24] — https://www.cdc.gov/sti/about/index.html
- See also: CDC clinical guidelines on the use of doxycycline postexposure prophylaxis for bacterial sexually transmitted infection prevention, United States, 2024 — http://dx.doi.org/10.15585/mmwr.rr7302a1